CLINICAL TRIAL: NCT04654793
Title: The Effect of Robotics-assisted Tilt Table and Functional Electrical Stimulation in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2017-0092
Record Dates: First submitted 2020-11-25; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Robot assisted inclined bed treatment and FES
  Interventions: Device: Robot assisted inclined bed treatment and FES
- Control group (Active Comparator): conventional inclined bed treatment
  Interventions: Device: conventional inclined bed treatment

INTERVENTIONS:
Device: Robot assisted inclined bed treatment and FES — FES was performed at the same time as the robot-assisted inclined bed treatment once a day for 30 minutes, 5 days a week for 4 weeks.
  Arms: Intervention group
Device: conventional inclined bed treatment — conventional inclined bed treatment for 30 minutes once a day for 4 weeks, 5 days a week
  Arms: Control group

SUMMARY:
Among subacute stroke patients (within 4 weeks after the onset), patients who are unable to walk are divided into experimental groups and control groups, and conventional rehabilitation treatment including physical therapy and occupational therapy is performed for 4 weeks or more in all groups.

Robot assisted inclined bed treatment and FES were performed, and the control group performed conventional inclined bed treatment.

The purpose of this study is to investigate the effect of robot-assisted inclined bed treatment by tracking observation and comparative analysis of the lower limb function, gait ability, bone density and muscle mass of each group.

Patients appropriate for the selection criteria are divided into experimental group and control group in random permuted blocks to conduct the study. In the experimental group, FES was performed at the same time as the robot-assisted inclined bed treatment once a day for 30 minutes, 5 days a week for 4 weeks, and the control group performed conventional inclined bed treatment for 30 minutes once a day for 4 weeks, 5 days a week. Separately from this in all groups, functional electrical stimulation treatment is performed once a day in the area except the lower extremities. In addition, all patients receive palliative physical therapy for 4 weeks for 1 hour a day. All subjects undergo a physical examination and whole body composition assessment before and after 4 weeks of treatment, and f/u after 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients within 4 weeks of onset of first stroke
2. Patients with an FAC score of 1 or less and at least one lower limb FMA of 15 or less
3. Adult male or female over 50 years of age
4. Those who have consented in writing to this clinical trial
5. A person who understands the purpose of the clinical trial and can adapt well to the treatment process

Exclusion Criteria:

1. Those with lower motor neuron lesions
2. A person who has an artificial implant due to a fracture of the lower extremity and spine, or a metal implant that generates an electrical signal such as an artificial pacemaker.
3. Those with a history of bone metabolism related diseases such as thyroid or parathyroid disease (excluding osteopenia and osteoporosis) or bone tumor
4. A person who has a history of fracture at the site of bone mineral density (ex. L1-L5, femoral head)
5. Those who have skin ulcers or skin diseases such as open wounds that make it difficult to apply robotic therapy
6. Those with the construction of the lower extremities
7. Those with deep vein thrombosis or arterial vascular disease of the lower extremities
8. Pregnant women
9. Not appropriate according to the judgment of other researchers

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-03-17 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment (lower) | before intervention
  A tool used to evaluate motor dysfunction, movement of the agonist and collaborator muscles, and coordination in stroke patients. It is used to evaluate motor function of the affected side.
Fugl-Meyer Assessment (lower) | 4weeks after
  A tool used to evaluate motor dysfunction, movement of the agonist and collaborator muscles, and coordination in stroke patients. It is used to evaluate motor function of the affected side.
Fugl-Meyer Assessment (lower) | 8weeks after
  A tool used to evaluate motor dysfunction, movement of the agonist and collaborator muscles, and coordination in stroke patients. It is used to evaluate motor function of the affected side.
Motricity Index | before intervention
  A tool used to evaluate motor power.
Motricity Index | 4weeks after
  A tool used to evaluate motor power.
Motricity Index | 8weeks after
  A tool used to evaluate motor power.
FAC (Functional ambulatory scale) | before intervention
  A tool to evaluate the independence of walking by measuring the degree of assistance required when walking. It is rated as 0-5 points.
FAC (Functional ambulatory scale) | 4weeks after
  A tool to evaluate the independence of walking by measuring the degree of assistance required when walking. It is rated as 0-5 points.
FAC (Functional ambulatory scale) | 8weeks after
  A tool to evaluate the independence of walking by measuring the degree of assistance required when walking. It is rated as 0-5 points.
Locomotion level of FIM (functional independence measure) | before intervention
  Indicator to evaluate independence in performing daily life movements
Locomotion level of FIM (functional independence measure) | 4weeks after
  Indicator to evaluate independence in performing daily life movements
Locomotion level of FIM (functional independence measure) | 8weeks after
  Indicator to evaluate independence in performing daily life movements
Berg balance scale | before intervention
  A tool to evaluate balance
Berg balance scale | 4weeks after
  A tool to evaluate balance
Berg balance scale | 8weeks after
  A tool to evaluate balance

CONTACTS AND LOCATIONS:
Overall Officials: Deog Young Kim, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No